CLINICAL TRIAL: NCT06116266
Title: NIDA CTN Protocol 0139: Collaborative Care for Polysubstance Use in Primary Care Settings (Co-Care)
Brief Title: Collaborative Care for Polysubstance Use in Primary Care Settings (Co-Care)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01169; UG1DA013035 (NIH)
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Educational Status; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-Care (Experimental): Patient participants with providers will receive primary care treatment plus the full Co-Care intervention which includes: Nurse Care Manager (NCM) visits, Addiction specialist consultations through NCM if indicated, and Health coaching sessions.
  Interventions: Other: Education and support for primary care providers (PCPS); Other: Nurse Care Manager (NCM) visits; Other: Addiction specialist consultant; Other: Health coaching sessions
- Enhanced Usual Care (EUC) (Active Comparator): Patient participants with providers will receive primary care treatment as usual plus educational materials.
  Interventions: Other: Education and support for primary care providers (PCPS); Other: Patient educational materials

INTERVENTIONS:
Other: Education and support for primary care providers (PCPS) — All PCPs in the EUC and Co-Care arms receive brief education on SUD treatment, including medications for OUD and AUD and contingency management for StUD, and recognizing and counteracting stigma while caring for patients with SUD.
Other: Nurse Care Manager (NCM) visits — A full-time clinic-embedded nurse care manager who works with patients and their PCPs to facilitate and support patient engagement in evidence-based treatment for polysubstance use and management of associated health conditions
  Arms: Co-Care
Other: Addiction specialist consultant — An addiction specialist consultant who supports the nurse care manager and PCP in formulating and adjusting treatment plans
  Arms: Co-Care
Other: Health coaching sessions — Health coaches who use motivational interviewing and cognitive behavioral therapy to motivate and support patients in behavior change to reduce polysubstance use-related harms. Patients may receive up to 12 health coaching sessions in total. The sessions will occur via phone and/or HIPAA compliant video chat software.
  Arms: Co-Care
Other: Patient educational materials — Patient participants receive an educational pamphlet addressing overdose prevention, information about accessing naloxone, and local SUD treatment options.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this trial is to test the efficacy of a collaborative care intervention to address opioid- and/or stimulant-involved polysubstance use in adult primary care patients with moderate to severe substance use disorders (SUD). The primary aims are to reduce days of opioid use (illicit or nonmedical opioid use), days of illicit stimulant use (cocaine, methamphetamine), and days of heavy alcohol use.

ELIGIBILITY:
PCP Inclusion Criteria:

* Licensed medical professional (MD, DO, NP, PA) who is able to prescribe controlled substances (Schedule III), or medical trainee meeting the requirements below.
* Serves as a primary care provider to adult patients (18 years of age and over) of the study clinic(s) during direct patient care sessions.
* Willing to be randomized to either of the study conditions. a. Medical trainees (physicians who are residents or fellows), are eligible if they have at least one continuity clinic session per week on average in the study clinic. Trainees must have plans to be working in a study clinic for approximately 8 months or longer. They must be able to provide prescriptions for controlled substances (Schedule III) either directly or through their preceptor(s).

Patient Inclusion Criteria:

* The participant's PCP is enrolled in the study.
* Age 18 years or older.
* Spoken and written proficiency in language of study materials, as determined by patient self-report and research staff evaluation.
* Moderate to severe substance use disorder for opioids, stimulants, and/or alcohol, (defined as meeting four or more DSM-5 criteria per substance as measured on the CIDI-adapted for DSM-5).
* a) Patients having alcohol use disorder without an opioid or stimulant SUD are required to have current opioid or stimulant use, as measured on the TAPS tool or baseline monthly survey.
* Current polysubstance use, defined as self-reported use of two or more substances of concern in the past 30 days, at least one of which is required to be an opioid or stimulant. Substances of concern include opioids (illicit opioids, nonmedical use of prescription opioids), stimulants (cocaine, methamphetamine), alcohol (heavy drinking defined as more than 5 for men and 4 for women drinks on a single occasion), and benzodiazepines (nonmedical use). Nonmedical use includes using prescription medications more than prescribed, or that were not prescribed to the individual taking them.
* Patients must report on the baseline monthly survey use in the past 30 days of at least one substance at or above the following thresholds: >10 days for opioids; >10 days for alcohol heavy drinking; >7 days for stimulants. These minimum thresholds reflect levels of use that are typical for individuals with moderate to severe SUD, and are lower for stimulants than for opioids and alcohol to reflect the different patterns of use that are observed in prior trials.
* Access to a reliable cell phone or willing to accept a phone as part of the incentive for completing the baseline visit (as determined by patient self-report).
* Able to provide sufficient contact information (minimum of one locator).
* Willing and able to provide written informed consent.

PCP Exclusion Criteria:

* Definite plan to resign from the clinic in the next eight months, per PCP self-report. Residents and fellows will need at least eight months before training completion to enroll.

Patient Exclusion Criteria:

* Currently being treated with medication for OUD (MOUD), and do not have moderate to severe AUD or StUD
* Initiated MOUD treatment (buprenorphine, methadone, or XR-NTX) within the 30 days prior to screening, per patient self-report. Because substance use may fall rapidly with the initiation of MOUD, patients who recently started MOUD may already be in the process of making changes to their substance use that are not attributable to the intervention.
* a) Initiation is defined as starting a new MOUD treatment episode, after not receiving MOUD treatment in the prior 30 days
* Initiated a SUD treatment program within the 30 days prior to screening, per patient self-report. Because substance use may fall rapidly with the initiation of a treatment program, patients who recently initiated treatment may already be making changes to their substance use that are not attributable to the intervention. SUD treatment program includes outpatient or residential programs for alcohol/drug treatment; does not include detox or short-term inpatient episodes (<15 days), or peer support (e.g., 12-Step Program such as AA/NA, Smart Recovery)
* a) Initiation is defined as starting a new treatment episode, after not being in a SUD treatment program in the prior 30 days
* Pregnancy, as determined by patient self-report.
* Are currently in jail, prison, or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities
* Definite plan to leave the area or the clinical practice within the next six months, per patient self-report.
* Other factors that may cause harm or increased risk to the participant or close contacts or preclude the patient's full adherence with or completion of the study (e.g. unstable/severe acute mental illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Total days of use of opioids, stimulants, and alcohol heavy drinking | Month 4-6
  Days of opioid use are defined as days with any use of heroin or synthetic opioids, or nonmedical use of prescription opioids. Nonmedical use includes using prescription opioids more than prescribed (e.g., taking two tablets when the prescription indicates a dose of one tablet) or taking pharmaceutical opioids that were not prescribed to the individual taking them. Days of stimulant use are defined as days with any use of cocaine or methamphetamine. Days of alcohol heavy drinking are defined as days with 5+ drinks/day for men, 4+ drinks/day for women.
  This outcome measure is collected using single item questions based on the Addiction Severity Index.
  Patient participants are asked to specify the number of days of use in the past 30 days (range is 0-30 days, value=0 for substances that were not used). The assessment is self-administered using a computerized form.

SECONDARY OUTCOMES:
Treatment Effectiveness Assessment (TEA) total score | Baseline
  The Treatment Effectiveness Assessment (TEA) is a 4-item patient-reported outcome measure of progress in treatment and recovery in the four following domains: substance use, health, lifestyle, and community involvement. Each domain is assessed with a single item and scored on a scale of 1-10 (higher scores indicate better progress). The total score is calculated using the sum of numerical responses for the four domains and can range from four (not well at all on all domains) to 40 (extremely well on all domains).
Treatment Effectiveness Assessment (TEA) total score | Month 3
  The Treatment Effectiveness Assessment (TEA) is a 4-item patient-reported outcome measure of progress in treatment and recovery in the four following domains: substance use, health, lifestyle, and community involvement. Each domain is assessed with a single item and scored on a scale of 1-10 (higher scores indicate better progress). The total score is calculated using the sum of numerical responses for the four domains and can range from four (not well at all on all domains) to 40 (extremely well on all domains).
Treatment Effectiveness Assessment (TEA) total score | Month 6
  The Treatment Effectiveness Assessment (TEA) is a 4-item patient-reported outcome measure of progress in treatment and recovery in the four following domains: substance use, health, lifestyle, and community involvement. Each domain is assessed with a single item and scored on a scale of 1-10 (higher scores indicate better progress). The total score is calculated using the sum of numerical responses for the four domains and can range from four (not well at all on all domains) to 40 (extremely well on all domains).
Treatment Effectiveness Assessment (TEA) total score | Month 12
  The Treatment Effectiveness Assessment (TEA) is a 4-item patient-reported outcome measure of progress in treatment and recovery in the four following domains: substance use, health, lifestyle, and community involvement. Each domain is assessed with a single item and scored on a scale of 1-10 (higher scores indicate better progress). The total score is calculated using the sum of numerical responses for the four domains and can range from four (not well at all on all domains) to 40 (extremely well on all domains).
Total days of use of opioids, stimulants, and alcohol | Months 10-12
  Days of opioid use are defined as days with any use of heroin or synthetic opioids, or nonmedical use of prescription opioids. Nonmedical use includes using prescription opioids more than prescribed (e.g., taking two tablets when the prescription indicates a dose of one tablet) or taking pharmaceutical opioids that were not prescribed to the individual taking them. Days of stimulant use are defined as days with any use of cocaine or methamphetamine. Days of alcohol heavy drinking are defined as days with 5+ drinks/day for men, 4+ drinks/day for women.
  This outcome measure is collected using single item questions based on the Addiction Severity Index. Patient participants are asked to specify the number of days of use in the past 30 days (range is 0-30 days, value=0 for substances that were not used). The assessment is self-administered using a computerized form.
Average days of abstinence from any unhealthy use of opioids, stimulants, and alcohol | Month 6
  Days of abstinence from substances of concern is measured as part of the Addiction Severity Index. At the end of the substance specific questions, patient participants who reported use of more than one substance of concern will be asked: "On how many days did you use none of these [insert names of all substances with 1+ days of use reported]?" (range is 0-30 days). For participants reporting use of 0-1 substances of concern, days of abstinence is calculated as 30 minus [number of days reported].
Average days of abstinence from any unhealthy use of opioids, stimulants, and alcohol | Month 12
  Days of abstinence from substances of concern is measured as part of the Addiction Severity Index. At the end of the substance specific questions, patient participants who reported use of more than one substance of concern will be asked: "On how many days did you use none of these [insert names of all substances with 1+ days of use reported]?" (range is 0-30 days). For participants reporting use of 0-1 substances of concern, days of abstinence is calculated as 30 minus [number of days reported].
Number of days of nonmedical benzodiazepine use | Baseline
  Nonmedical benzodiazepine use is defined as taking benzodiazepines that were not prescribed to the individual taking them.
  This outcome measure will be measured using single item questions based on the Addiction Severity Index. "During the past 30 days, on how many days did you use [substance name]?" The question will be asked separately for each substance type. Patient participants are asked to specify the number of days of use in the past 30 days (range is 0-30 days, value=0 for substances that were not used). The assessment is self-administered using a computerized form.
Number of days of nonmedical benzodiazepine use | Months 4-6
  Nonmedical benzodiazepine use is defined as taking benzodiazepines that were not prescribed to the individual taking them.
  This outcome measure will be measured using single item questions based on the Addiction Severity Index. "During the past 30 days, on how many days did you use [substance name]?" The question will be asked separately for each substance type. Patient participants are asked to specify the number of days of use in the past 30 days (range is 0-30 days, value=0 for substances that were not used). The assessment is self-administered using a computerized form.
Number of days of nonmedical benzodiazepine use | Months 10-12
  Nonmedical benzodiazepine use is defined as taking benzodiazepines that were not prescribed to the individual taking them.
  This outcome measure will be measured using single item questions based on the Addiction Severity Index. "During the past 30 days, on how many days did you use [substance name]?" The question will be asked separately for each substance type. Patient participants are asked to specify the number of days of use in the past 30 days (range is 0-30 days, value=0 for substances that were not used). The assessment is self-administered using a computerized form.
Proportion of patients with receipt of a prescription for a medication used for SUD treatment | Baseline
  Medication for SUD is defined as any medication for OUD, AUD, or StUD. This measures is collected from the electronic health record.
Proportion of patients with receipt of a prescription for a medication used for SUD treatment | Month 3
  Medication for SUD is defined as any medication for OUD, AUD, or StUD. This measures is collected from the electronic health record.
Proportion of patients with receipt of a prescription for a medication used for SUD treatment | Month 6
  Medication for SUD is defined as any medication for OUD, AUD, or StUD. This measures is collected from the electronic health record.
Proportion of patients with receipt of a prescription for a medication used for SUD treatment | Month 12
  Medication for SUD is defined as any medication for OUD, AUD, or StUD. This measures is collected from the electronic health record.
Proportion of patients attending behavioral health visit(s) addressing substance use | Baseline
  This measure is based on behavioral health visits addressing substance use that occurred in the study clinic(s), as documented in the electronic health record.
Proportion of patients attending behavioral health visit(s) addressing substance use | Month 3
  This measure is based on behavioral health visits addressing substance use that occurred in the study clinic(s), as documented in the electronic health record.
Proportion of patients attending behavioral health visit(s) addressing substance use | Month 6
  This measure is based on behavioral health visits addressing substance use that occurred in the study clinic(s), as documented in the electronic health record.
Proportion of patients attending behavioral health visit(s) addressing substance use | Month 12
  This measure is based on behavioral health visits addressing substance use that occurred in the study clinic(s), as documented in the electronic health record.
OUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Baseline
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The OUD category in the questionnaire is comprised of 15 yes/no items. The OUD symptom score is calculated by finding the sum of the items marked "Yes". OUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
OUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Month 6
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The OUD category in the questionnaire is comprised of 15 yes/no items. The OUD symptom score is calculated by finding the sum of the items marked "Yes". OUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
StUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Baseline
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The StUD category in the questionnaire is comprised of 15 yes/no items. The StUD symptom score is calculated by finding the sum of the items marked "Yes". StUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
StUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Month 6
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The StUD category in the questionnaire is comprised of 15 yes/no items. The StUD symptom score is calculated by finding the sum of the items marked "Yes". StUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
AUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Baseline
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The AUD category in the questionnaire is comprised of 15 yes/no items. The AUD symptom score is calculated by finding the sum of the items marked "Yes". AUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
AUD symptom score from the Modified World Mental Health Composite International Diagnostic Interview (CIDI) questionnaire | Month 6
  The CIDI questionnaire measures severity of symptoms for three categories of substance use disorders (SUD); OUD, StUD, and AUD. The AUD category in the questionnaire is comprised of 15 yes/no items. The AUD symptom score is calculated by finding the sum of the items marked "Yes". AUD scores are interpreted as follows: 0-1 (subthreshold), 2-3 (mild use disorder), 4-5 (moderate use disorder), and 6+ (severe use disorder).
Overdose Risk Behavior Questionnaire score | Baseline
  The Overdose Risk Behavior Questionnaire is a 9-item self-administered questionnaire. These questions measure the frequency, in the past 6 months, at which individuals used alone; used in a new place/environment; used other substances (alcohol, benzodiazepines, stimulants) within 2 hours of opioids; used more than one opioid; used more than the usual amount; and used inhaled or injected opioids. Response options were "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)," except for #6, which was "never (0)," "once (1)," or "more than once (2)." The total risk score is an aggregation of responses to the individual questions. Sum score range: 0-32, higher scores indicate greater risk of overdose.
Overdose Risk Behavior Questionnaire score | Month 6
  The Overdose Risk Behavior Questionnaire is a 9-item self-administered questionnaire. These questions measure the frequency, in the past 6 months, at which individuals used alone; used in a new place/environment; used other substances (alcohol, benzodiazepines, stimulants) within 2 hours of opioids; used more than one opioid; used more than the usual amount; and used inhaled or injected opioids. Response options were "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)," except for #6, which was "never (0)," "once (1)," or "more than once (2)." The total risk score is an aggregation of responses to the individual questions. Sum score range: 0-32, higher scores indicate greater risk of overdose.
Overdose Risk Behavior Questionnaire score | Month 12
  The Overdose Risk Behavior Questionnaire is a 9-item self-administered questionnaire. These questions measure the frequency, in the past 6 months, at which individuals used alone; used in a new place/environment; used other substances (alcohol, benzodiazepines, stimulants) within 2 hours of opioids; used more than one opioid; used more than the usual amount; and used inhaled or injected opioids. Response options were "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)," except for #6, which was "never (0)," "once (1)," or "more than once (2)." The total risk score is an aggregation of responses to the individual questions. Sum score range: 0-32, higher scores indicate greater risk of overdose.
Number of episodes of a non-fatal overdose | Baseline
  Outcome measure is self reported on the Non-Fatal Overdose Questionnaire.
Number of episodes of a non-fatal overdose | Month 6
  Outcome measure is self reported on the Non-Fatal Overdose Questionnaire.
Number of episodes of a non-fatal overdose | Month 12
  Outcome measure is self reported on the Non-Fatal Overdose Questionnaire.
World Health Organization Quality of Life (WHOQOL-BREF) score | Baseline
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. The mean score of items within each domain is used to calculate the domain score. After computed the scores, they transformed linearly to a 0-100-scale. Higher scores denote higher QOL.
World Health Organization Quality of Life (WHOQOL-BREF) score | Month 3
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. The mean score of items within each domain is used to calculate the domain score. After computed the scores, they transformed linearly to a 0-100-scale. Higher scores denote higher QOL.
World Health Organization Quality of Life (WHOQOL-BREF) score | Month 6
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. The mean score of items within each domain is used to calculate the domain score. After computed the scores, they transformed linearly to a 0-100-scale. Higher scores denote higher QOL.
World Health Organization Quality of Life (WHOQOL-BREF) score | Month 12
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. The mean score of items within each domain is used to calculate the domain score. After computed the scores, they transformed linearly to a 0-100-scale. Higher scores denote higher QOL.
Single-item general health question (HRQOL-1) score | Baseline
  Questionnaire consist of one question 'Would you say that in general your health is' [scaled response ranges from (5)Excellent, (4)Very good, (3)Good, (2)Fair or (1)Poor]. The higher the score the better the patient's general health.
Single-item general health question (HRQOL-1) score | Month 3
  Questionnaire consist of one question 'Would you say that in general your health is' [scaled response ranges from (5)Excellent, (4)Very good, (3)Good, (2)Fair or (1)Poor]. The higher the score the better the patient's general health.
Single-item general health question (HRQOL-1) score | Month 6
  Questionnaire consist of one question 'Would you say that in general your health is' [scaled response ranges from (5)Excellent, (4)Very good, (3)Good, (2)Fair or (1)Poor]. The higher the score the better the patient's general health.
Single-item general health question (HRQOL-1) score | Month 12
  Questionnaire consist of one question 'Would you say that in general your health is' [scaled response ranges from (5)Excellent, (4)Very good, (3)Good, (2)Fair or (1)Poor]. The higher the score the better the patient's general health.
Patient Health Questionnaire (PHQ-8) score | Baseline
  The Patient Health Questionnaire depression scale (PHQ-8) consists of 8 items. The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Patient Health Questionnaire (PHQ-8) score | Month 3
  The Patient Health Questionnaire depression scale (PHQ-8) consists of 8 items. The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Patient Health Questionnaire (PHQ-8) score | Month 6
  The Patient Health Questionnaire depression scale (PHQ-8) consists of 8 items. The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Patient Health Questionnaire (PHQ-8) score | Month 12
  The Patient Health Questionnaire depression scale (PHQ-8) consists of 8 items. The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Percentage of participants with a negative suicidality screen | Baseline
  Outcome measured by Ask Suicide-Screening Questions (ASQ). The ASQ consists of four yes/no questions. If patient answers "No" to all questions 1 through 4, they are considered negative for suicidality. If patient answers "Yes" to any of questions 1 through 4, or refuses to answer, they are considered a positive screen.
Percentage of participants with a negative suicidality screen | Month 3
  Outcome measured by Ask Suicide-Screening Questions (ASQ). The ASQ consists of four yes/no questions. If patient answers "No" to all questions 1 through 4, they are considered negative for suicidality. If patient answers "Yes" to any of questions 1 through 4, or refuses to answer, they are considered a positive screen.
Percentage of participants with a negative suicidality screen | Month 6
  Outcome measured by Ask Suicide-Screening Questions (ASQ). The ASQ consists of four yes/no questions. If patient answers "No" to all questions 1 through 4, they are considered negative for suicidality. If patient answers "Yes" to any of questions 1 through 4, or refuses to answer, they are considered a positive screen.
Percentage of participants with a negative suicidality screen | Month 12
  Outcome measured by Ask Suicide-Screening Questions (ASQ). The ASQ consists of four yes/no questions. If patient answers "No" to all questions 1 through 4, they are considered negative for suicidality. If patient answers "Yes" to any of questions 1 through 4, or refuses to answer, they are considered a positive screen.
Generalized Anxiety Disorder (GAD-7) score | Baseline
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The whole scale score can range from 0 to 21 Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Generalized Anxiety Disorder (GAD-7) score | Month 3
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The whole scale score can range from 0 to 21 Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Generalized Anxiety Disorder (GAD-7) score | Month 6
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The whole scale score can range from 0 to 21 Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Generalized Anxiety Disorder (GAD-7) score | Month 12
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The whole scale score can range from 0 to 21 Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Primary Care Post-Traumatic Disorder Screen for DSM-5 (PC-PTSD-5) score | Baseline
  PC-PTSD-5 consists of 5-items. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0 meaning no trauma exposure. If a respondent endorses a trauma exposure, they can score a 0-5 on the PC-PTSD-5, which is a count of "yes" responses to the 5 questions about how the trauma has affected them in the past month. Higher scores indicate the trauma exposure has often affected them over the past month.
Primary Care Post-Traumatic Disorder Screen for DSM-5 (PC-PTSD-5) score | Month 3
  PC-PTSD-5 consists of 5-items. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0 meaning no trauma exposure. If a respondent endorses a trauma exposure, they can score a 0-5 on the PC-PTSD-5, which is a count of "yes" responses to the 5 questions about how the trauma has affected them in the past month. Higher scores indicate the trauma exposure has often affected them over the past month.
Primary Care Post-Traumatic Disorder Screen for DSM-5 (PC-PTSD-5) score | Month 6
  PC-PTSD-5 consists of 5-items. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0 meaning no trauma exposure. If a respondent endorses a trauma exposure, they can score a 0-5 on the PC-PTSD-5, which is a count of "yes" responses to the 5 questions about how the trauma has affected them in the past month. Higher scores indicate the trauma exposure has often affected them over the past month.
Primary Care Post-Traumatic Disorder Screen for DSM-5 (PC-PTSD-5) score | Month 12
  PC-PTSD-5 consists of 5-items. If a respondent denies exposure, the PC-PTSD-5 is complete with a score of 0 meaning no trauma exposure. If a respondent endorses a trauma exposure, they can score a 0-5 on the PC-PTSD-5, which is a count of "yes" responses to the 5 questions about how the trauma has affected them in the past month. Higher scores indicate the trauma exposure has often affected them over the past month.
Number of Patient Reported ED visits | Baseline
Number of Patient Reported ED visits | Month 6
Number of Patient Reported ED visits | Month 12
Number of patient reported hospital admissions | Baseline
Number of patient reported hospital admissions | Month 6
Number of patient reported hospital admissions | Month 12
Proportion of patients with a diagnosis of OUD receiving any medication for OUD treatment | Month 12
Proportion of patients with a diagnosis of AUD receiving any medication for AUD treatment | Month 12
PCPs Medical Condition Regard Scale (MCRS) score | Baseline
  Medical Condition Regard Scale (MCRS) is a self-administered instrument examines the degree to which 12 medical conditions (including alcohol dependence and intravenous drug use) are enjoyable, treatable, and worthy of medical resources. Responses were measured on a six-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = not sure but probably disagree, 4 = not sure but probably agree, 5 = agree, and 6 = strongly agree. A MCRS score of >57 correlates with high probability of desire to care for patients with with drug and alcohol use.
PCPs Medical Condition Regard Scale (MCRS) score | End of intervention period, up to 21 months
  Medical Condition Regard Scale (MCRS) is a self-administered instrument examines the degree to which 12 medical conditions (including alcohol dependence and intravenous drug use) are enjoyable, treatable, and worthy of medical resources. Responses were measured on a six-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = not sure but probably disagree, 4 = not sure but probably agree, 5 = agree, and 6 = strongly agree. A MCRS score of >57 correlates with high probability of desire to care for patients with with drug and alcohol use.
PCPs REDUCE-HARM instrument score | Baseline
  The REDUCE-HARM instrument is a 24-item scale to measure healthcare professional attitudes to work with people who inject drugs including self-reported skills in different aspects of substance use as well as attitudes towards individuals who use drugs. Each item is ranked from 1 = not at all important to 3 = very important. Higher scores indicate positive attitudes toward caring for patients with SUD.
PCPs REDUCE-HARM instrument score | End of intervention period, up to 21 months
  The REDUCE-HARM instrument is a 24-item scale to measure healthcare professional attitudes to work with people who inject drugs including self-reported skills in different aspects of substance use as well as attitudes towards individuals who use drugs. Each item is ranked from 1 = not at all important to 3 = very important. Higher scores indicate positive attitudes toward caring for patients with SUD.
PCPs Addictions Knowledge Questions score | Baseline
  The Addictions Knowledge Questions is a 6-question measure that asks basic knowledge questions about DSM-criteria for SUD, and pharmacological treatments for OUD and AUD. Each item is answered by the PCP with a choice of "Correct" or "Incorrect". The score is calculated by the adding the number of items that are answered with "Correct". Total scores range from 0-6, a higher score indicating better knowledge.
PCPs Addictions Knowledge Questions score | End of intervention period, up to 21 months
  The Addictions Knowledge Questions is a 6-question measure that asks basic knowledge questions about DSM-criteria for SUD, and pharmacological treatments for OUD and AUD. Each item is answered by the PCP with a choice of "Correct" or "Incorrect". The score is calculated by the adding the number of items that are answered with "Correct". Total scores range from 0-6, a higher score indicating better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, MD, Principal Investigator — NYU Langone Health
Locations (8):
- United States (8):
  - Harbor-UCLA Medical Center, Torrance, California
  - NYU Langone Health, New York, New York
  - The Institute for Family Health, New York, New York
  - Winding Waters Medical Clinic, Enterprise, Oregon
  - Union Community Care, Lancaster, Pennsylvania
  - Harris Health, Houston, Texas
  - Sea Mar Community Health Centers, Bellingham, Washington
  - Wisconsin Research & Education Network, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Implementation Guidance (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm) and (for HEAL-funded studies) the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy).
  Primary data for this study will be available to the public in the NIDA data repository. For more details on data sharing please visit https://datashare.nida.nih.gov/.
  The primary outcome(s) publication will be included along with study underlying primary data in the data share repository, and it will also be deposited in PubMed Central http://www.pubmedcentral.nih.gov/ per NIH Policy (http://publicaccess.nih.gov/).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Anyone who wishes to access the data for any purpose can find that data is available indefinitely at (https://datashare.nida.nih.gov/).
URL: https://datashare.nida.nih.gov/